CLINICAL TRIAL: NCT04378972
Title: Analysis of Soluble Mediators of Inflammation and Angiogenesis in the Vitreous of Patients With Diabetic Retinopathy Treated With Curcumin/Homotaurine/Vit. D3
Brief Title: Anti-inflammatory Effect of Curcumin, Homotaurine, Vitamin D3 on Human Vitreous in Patients With Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: University of Molise (Other)
Collaborators: Humanitas Gradenigo - Torino (Unknown); Cliniche Humanitas Gavazzeni (Other); Consorzio Sannio Tech (Other); University of Roma La Sapienza (Other); FB VISION, Ascoli Piceno, Italy (Unknown)
Responsible Party: Principal Investigator, Ciro Costagliola, Full Professor in Ophthalmology, University of Molise
Other Study IDs: 11/2019
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Diabetic Retinopathy
Keywords: neuroprotection; vitreous; pro-inflammatory cytokines; curcumin; vitamin D3; homotaurine
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Curcumin; tramiprosate; Cholecalciferol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — human vitreous
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TREATED GROUP: 25 portions of vitreous samples from 25 eyes of patients operated on vitrectomy for complications from diabetic retinopathy, incubated with curcumin, homotaurine and vitamin D3. The substances will be used individually and in triple association, to evaluate a possible synergistic effect on the expression of inflammatory cytokines and endothelial growth factors.
  Interventions: Other: curcumin, homotaurine, vitamin D3
- CONTROL GROUP: The same fractions of vitreous samples (n = 25) evaluated for the expression of oxidative biomarkers, inflammatory cytokines and metalloproteinases, without prior incubation with the substances of the treated group.
  Interventions: Other: control

INTERVENTIONS:
Other: curcumin, homotaurine, vitamin D3 — ELISA tests on supernatants of 25 vitreous biopsies incubated with bioactive molecules at 37 ° C for 20 h. The concentration of soluble mediators was calculated from a calibration curve.
  Groups: TREATED GROUP
Other: control — ELISA tests on supernatants of 25 vitreous biopsies. The concentration of soluble mediators was calculated from a calibration curve.
  Groups: CONTROL GROUP

SUMMARY:
Dosage of pro-inflammatory cytokines and soluble mediators (TNFα, IL6, IL2 and PDGF-AB) performed on 25 vitreous biopsies taken from patients with diabetic retinopathy and treated with increasing doses of curcumin (0.5uM and 1uM), with or without homotaurine (100uM) and vitamin D3 (50nM).

DETAILED DESCRIPTION:
Diabetic retinopathy is one of the most common complications of diabetes mellitus and is a leading cause of vision loss and blindness in the working-age population worldwide. DR is being recognized as a neurodegenerative disease of the retina as opposed to previously considered solely as a microvascular disease. Progressive blindness is due to the long-term accumulation of pathological abnormalities in the retina of hyperglycemic patients. In the initial phase, non-proliferative diabetic retinopathy (NPDR) is almost asymptomatic with the onset of microhemorrhagic and microischemic episodes and an increase in vascular permeability. Subsequently, the progression of the disease is accompanied by the onset of a chronic inflammatory state and neovascularization in a vicious circle that feeds and determines the accumulation of damage to the retina through hypoxia, oxidative stress and widespread neurodegeneration. Among metabolites, hyperglycemia is known to be the major factor which activates several metabolic pathways harmful for retina. Moreover, an increased level of glutamate has been reported in the diabetic retina and also in the vitreous of diabetic patients, suggesting a neurotoxic role of glutamate which may damage retinal neurons and especially retinal ganglion cells by excitotoxicity. In proliferative diabetic retinopathy (PDR), vitreous humor undergoes structural and molecular changes, with changes also in composition, which play a central role in supporting disease progression.The vitreous, 4 ml in volume, is a transparent gel-like structure which fills the space between the lens and the retina. It is composed of 98-99% of water with traces of cations, ions, proteins (mainly collagen) and polysaccharides such as hyaluronic acid. In PDR patients undergoing pars plana vitrectomy, vitreous samples are characterized by altered levels of bioactive molecules with pro-angiogenic, proinflammatory and neuromodulatory activities. So, it is clear that the vitreous acts as a reservoir of soluble signaling mediators that could exacerbate retinal damage. On the other hand, the vitreous obtained from patients with PDR can be a powerful tool to evaluate the anti-angiogenic / anti-inflammatory activity of new biomolecules that could be potential candidates for the treatment of diabetic vitreoretinopathy. Currently, PDR is treated with laser photocoagulation, vitreoretinal surgery or intravitreal injection of drugs targeted to the vascular endothelial growth factor (VEGF) and steroid agents.However, these protocols are effective in the short term, cause side effects and, above all, are indicated only for advanced stages of the disease. So, noninvasive, nondestructive, and longer-duration treatment options are also needed. Recently, research eﬀorts have been made to identify neuroprotective drugs able to prevent visual ﬁeld loss and preserve visual function and a promising alternative for the treatment of early-stage NPDR comes from nutraceuticals. In fact, in vitro and in vivo studies have revealed that a variety of nutraceuticals has important antioxidant and anti-inflammatory properties that can compromise the first diabetes-driven molecular events that cause vitreoretinopathy, acting upstream of the disease. Based on the results of several investigations, it is reasonable to assert that a single constituent that aﬀects one target has limited eﬃcacy in preventing the progression of multifactorial diseases. A large body of research revealed that the use of a combination of compounds with synergistic multitarget eﬀects may oﬀer a more powerful approach for disease prevention, including retinal neurodegeneration. In experimental models of retinal neurodegeneration it has been shown that cotreatment of citicoline and homotaurine has a direct neuroprotective eﬀect on primary retinal cells exposed to glutamate toxicity and HG levels. Glutamate-induced excitotoxicity is implicated in the pathophysiology of several degenerative diseases of the retina, including glaucoma. Moreover, HG-induced neurotoxicity is a characteristic of diabetic retinopathy. Curcumin, a yellowish non-flavonoid polyphenol that constitutes the main active compound of Curcuma longa, is widely known for its antioxidant and anti-inflammatory properties . Many studies have also described its marked protective effect on retinal cells against oxidative stress and inflammation. Lastly, vitamin D levels appeared to be lower in diabetes mellitus type 2 patients and this could have therapeutic implications. Therefore, the aim of the investigator's study is to analyze the soluble mediators of inflammation and angiogenesis in the vitreous of patients with diabetic retinopathy treated with homotaurine, curcumin and vitamin D3.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* patients with diabetic retinopathy requiring vitrectomy
* willingness to participate in the study following its indications

Exclusion Criteria:

* previous vitrectomy in the study eye
* previous buckle surgery in the study eye
* previous intravitreal injection in the study eye
* concurrent retinovascular or other ocular inflammatory disease
* history of ocular trauma
* concomitant intake of any topical or systemic NSAID or corticosteroid therapy
* presence of systemic inflammations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 patients aged ≥18 years with diabetic retinopathy requiring vitrectomy
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-11-16 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
pro-inflammatory cytokines analysis | 7 days
  Evaluation of the anti-inflammatory effect of curcumin, homotaurine and vitamin D3 on the expression of inflammatory cytokines in human vitreous samples of patients suffering from diabetic retinopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Costagliola, Full Professor, Principal Investigator — University of Molise
Locations (1):
- University of Molise, Campobasso, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stefansson E, Bek T, Porta M, Larsen N, Kristinsson JK, Agardh E. Screening and prevention of diabetic blindness. Acta Ophthalmol Scand. 2000 Aug;78(4):374-85. doi: 10.1034/j.1600-0420.2000.078004374.x. PMID 10990036
- [Result] Bringmann A, Iandiev I, Pannicke T, Wurm A, Hollborn M, Wiedemann P, Osborne NN, Reichenbach A. Cellular signaling and factors involved in Muller cell gliosis: neuroprotective and detrimental effects. Prog Retin Eye Res. 2009 Nov;28(6):423-51. doi: 10.1016/j.preteyeres.2009.07.001. Epub 2009 Aug 4. PMID 19660572
- [Result] Cheung N, Mitchell P, Wong TY. Diabetic retinopathy. Lancet. 2010 Jul 10;376(9735):124-36. doi: 10.1016/S0140-6736(09)62124-3. Epub 2010 Jun 26. PMID 20580421
- [Result] Antonetti DA, Klein R, Gardner TW. Diabetic retinopathy. N Engl J Med. 2012 Mar 29;366(13):1227-39. doi: 10.1056/NEJMra1005073. No abstract available. PMID 22455417
- [Result] Bringmann A, Wiedemann P. Muller glial cells in retinal disease. Ophthalmologica. 2012;227(1):1-19. doi: 10.1159/000328979. Epub 2011 Sep 15. PMID 21921569
- [Result] El-Asrar AM. Role of inflammation in the pathogenesis of diabetic retinopathy. Middle East Afr J Ophthalmol. 2012 Jan;19(1):70-4. doi: 10.4103/0974-9233.92118. PMID 22346117
- [Result] Morescalchi F, Duse S, Gambicorti E, Romano MR, Costagliola C, Semeraro F. Proliferative vitreoretinopathy after eye injuries: an overexpression of growth factors and cytokines leading to a retinal keloid. Mediators Inflamm. 2013;2013:269787. doi: 10.1155/2013/269787. Epub 2013 Sep 30. PMID 24198445
- [Result] dell'Omo R, Semeraro F, Bamonte G, Cifariello F, Romano MR, Costagliola C. Vitreous mediators in retinal hypoxic diseases. Mediators Inflamm. 2013;2013:935301. doi: 10.1155/2013/935301. Epub 2013 Jan 10. PMID 23365490
- [Result] Wu L, Fernandez-Loaiza P, Sauma J, Hernandez-Bogantes E, Masis M. Classification of diabetic retinopathy and diabetic macular edema. World J Diabetes. 2013 Dec 15;4(6):290-4. doi: 10.4239/wjd.v4.i6.290. PMID 24379919
- [Result] Cunha-Vaz J, Ribeiro L, Lobo C. Phenotypes and biomarkers of diabetic retinopathy. Prog Retin Eye Res. 2014 Jul;41:90-111. doi: 10.1016/j.preteyeres.2014.03.003. Epub 2014 Mar 26. PMID 24680929
- [Result] Grigsby JG, Cardona SM, Pouw CE, Muniz A, Mendiola AS, Tsin AT, Allen DM, Cardona AE. The role of microglia in diabetic retinopathy. J Ophthalmol. 2014;2014:705783. doi: 10.1155/2014/705783. Epub 2014 Aug 31. PMID 25258680
- [Result] Jenkins AJ, Joglekar MV, Hardikar AA, Keech AC, O'Neal DN, Januszewski AS. Biomarkers in Diabetic Retinopathy. Rev Diabet Stud. 2015 Spring-Summer;12(1-2):159-95. doi: 10.1900/RDS.2015.12.159. Epub 2015 Aug 10. PMID 26676667
- [Result] Semeraro F, Cancarini A, dell'Omo R, Rezzola S, Romano MR, Costagliola C. Diabetic Retinopathy: Vascular and Inflammatory Disease. J Diabetes Res. 2015;2015:582060. doi: 10.1155/2015/582060. Epub 2015 Jun 7. PMID 26137497
- [Result] Semeraro F, Russo A, Gambicorti E, Duse S, Morescalchi F, Vezzoli S, Costagliola C. Efficacy and vitreous levels of topical NSAIDs. Expert Opin Drug Deliv. 2015;12(11):1767-82. doi: 10.1517/17425247.2015.1068756. Epub 2015 Jul 14. PMID 26173446
- [Result] Bolinger MT, Antonetti DA. Moving Past Anti-VEGF: Novel Therapies for Treating Diabetic Retinopathy. Int J Mol Sci. 2016 Sep 7;17(9):1498. doi: 10.3390/ijms17091498. PMID 27618014
- [Result] Nawaz IM, Rezzola S, Cancarini A, Russo A, Costagliola C, Semeraro F, Presta M. Human vitreous in proliferative diabetic retinopathy: Characterization and translational implications. Prog Retin Eye Res. 2019 Sep;72:100756. doi: 10.1016/j.preteyeres.2019.03.002. Epub 2019 Apr 2. PMID 30951889
- [Derived] Filippelli M, Campagna G, Vito P, Zotti T, Ventre L, Rinaldi M, Bartollino S, dell'Omo R, Costagliola C. Anti-inflammatory Effect of Curcumin, Homotaurine, and Vitamin D3 on Human Vitreous in Patients With Diabetic Retinopathy. Front Neurol. 2021 Feb 5;11:592274. doi: 10.3389/fneur.2020.592274. eCollection 2020. PMID 33633656